CLINICAL TRIAL: NCT03817554
Title: A Randomized Controlled Trial of Pramipexole for Restless Leg Syndrome in Peritoneal Dialysis Patients
Brief Title: Pramipexole for Restless Leg Syndrome in Peritoneal Dialysis Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The recruitment of participants in the study was difficulty.
Sponsor: Dong Jie (Other)
Responsible Party: Sponsor-Investigator, Dong Jie, Clinical Professor, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pramipexole
Record Dates: First submitted 2019-01-11; First posted 2019-01-25 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Restless Legs Syndrome
Keywords: Pramipexole,; Restless Leg Syndrome; Peritoneal Dialysis
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole; Dopamine Agonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment group (Experimental): Peritoneal dialysis patients diagnosed with restless legs syndrome will receive pramipexole.
  Interventions: Drug: Pramipexole; Other: placebo
- Control group (Placebo Comparator): Peritoneal dialysis patients diagnosed with restless legs syndrome will receive placebo.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Pramipexole — Pramipexole will be taken once daily in the evening 2 to 3 hours before bedtime. The starting dose of pramipexole is 0.125 mg/day. During the first 4 weeks, the daily dose could be increased by the treating physician in weekly intervals to 0.25, 0.50, or 0.75 mg/day, according to the Patient Global Impression scale (PGI) rating and overall tolerability of the drug. In the case of adverse events (AEs), the dose could be reduced to the previous dose step. During 5 to 12 weeks, the dose will keep constant.
  Other Names: Dopamine Agonist
  Arms: Treatment group
Other: placebo — Placebo will be taken once daily in the evening 2 to 3 hours before bedtime. The starting dose of placebo is 0.125 mg/day. During the first 4 weeks, the daily dose could be increased by the treating physician in weekly intervals to 0.25, 0.50, or 0.75 mg/day, according to the Patient Global Impression scale (PGI) rating and overall tolerability of the drug. In the case of adverse events (AEs), the dose could be reduced to the previous dose step. During 5 to 12 weeks, the dose will keep constant.

SUMMARY:
A randomized, double-blind controlled Study from a single center to evaluate the effect and safety of pramipexole on peritoneal dialysis patients with restless legs syndrome

DETAILED DESCRIPTION:
Peritoneal dialysis patients diagnosed with restless legs syndrome will be divided into experiment group and control group, and will be prescribed with pramipexole and placebo respectively.After 12 weeks, we will compare IRLSSG（International RLS Study Group Rating Scale）、MOS（Medical Outcomes Study ）Sleeping Scale、Self-Rating Anxiety Scale and Self-Rating Depression Scale before and after the prescription.

ELIGIBILITY:
Inclusion Criteria:

1. PD patients (aged ≥18 years) are dialyzed with lactate-buffered glucose dialysate, using a twinbag connection system (Baxter Healthcare, Guangzhou, China).
2. For entry , all patients are required to meet all diagnositic criteria of the International RLS Study Group (IRLSSG), to have a baseline total score >15 on the Study Group's International RLS Rating Scale (IRLS), and to have experienced RLS symptoms at least 2-3 days per week throughout the perior 3 months.
3. Each patient should write informed consent.
4. All patients are required to be interviewed to the frequency required by the research process.

Exclusion Criteria:

1. Patients with severe gastrointestinal illness can not tolerate oral drugs.
2. Patients who work on a shift schedule are not allowed to participate.
3. Women with childbearing potential are excluded for pregnancy, inadequate contraception, or current breastfeeding of a child.
4. Patients are also excluded for current use (within 14 days before baseline) of medications that might affect RLS symptoms, e.g., levodopa, dopamine agonists or antagonists, hypnotics, lithium formulations, or antidepressants.
5. Patients with serum ferritin ≤200 ng/ml, or Hb <110g/L, or Kt/V <1.7 are excluded.
6. Patients with severe and unstable inflammation disease (active systemic infection, acute cardiovascular disease, active liver disease, active connective tissue disorder, ,and cancer within 1 year of radiotherapy and chemotherapy, )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Absolute change in IRLSSG Score | 12 weeks
  Absolute change in IRLS sum score will be defined as a change in IRLSSG from baseline to the end of treatment phase. The scale range from 0 to 40. The higher values represent a worse outcome.

SECONDARY OUTCOMES:
Effect on Sleep assessment Questionnaire | 12 weeks
  The absolute change of Sleep assessment Questionnaire between baseline and the twelfth week.The scale range from 0 to 60. The higher values represent a worse outcome.
Effect on Quality of life (QoL) questionare | 12 weeks
  The absolute change of QoL between baseline and the twelfth week. The scale range from 20 to 60. The higher values represent a worse outcome.The scale range from 36 to 162. The higher values represent a worse outcome.
Effect on self rating anxiety scale | 12 weeks
  The absolute change of self rating anxiety between baseline and the twelfth week. The scale range from 35 to 85. The higher values represent a worse outcome.
Effect on depression self rating scale | 12 weeks
  The absolute change of depression self rating between baseline and the twelfth week. The absolute change of self rating anxiety between baseline and the twelfth week. The scale range from 20 to 60. The higher values represent a worse outcome.
Effects on Blood pressure | 12 weeks
  The absolute change of 24-hour ambulatory blood pressure monitoring between baseline and the twelfth week. Both systolic and diastolic pressures will be assessed during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, Study Director — Peking Universiy First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma TT, Yang Z, Zhu S, Zhao JH, Li Y, Sun FY, Zhao N, Xiong ZY, Xiong ZB, Dong J. Pramipexole in peritoneal dialysis patients with restless legs syndrome (RLS): a protocol for a multicentre double-blind randomised controlled trial. BMJ Open. 2020 Feb 18;10(2):e033815. doi: 10.1136/bmjopen-2019-033815. PMID 32075834